CLINICAL TRIAL: NCT04016883
Title: Effect of Problem-solving Therapy Offered Through a Web Platform on Levels of Perceived Stress by Administrative Workers: A Controlled Randomized Trial
Brief Title: Effect of Problem-solving Therapy Offered Through a Web Platform on Levels of Stress
Acronym: PST on stress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Katherine Linda Arapa Apaza, Researcher, Universidad Peruana Cayetano Heredia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 103876
Record Dates: First submitted 2019-07-08; First posted 2019-07-12 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Stress, Psychological; Behavior; Occupational Stress; Mental Health Wellness 1
MeSH Terms: conditions — Stress, Psychological; Behavior; Occupational Stress

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled trial of parallel type (2 arms, with a ratio of 1: 1, and with a block size of 5), which consists of the following phases where necessary changes in the methods are described after to start the trial:
Who Masked: Investigator
Masking Description: double-blind masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional web platform (Sham Comparator): Participants asked to review the web platform for 4 weeks.
  Interventions: Other: Conventional web platform
- Problem Solving Therapy offered through a web platform (Experimental): 4 sessions with cognitive behavioral therapy, offered through a web platform. Each session will be offered per week.
  Interventions: Other: Problem Solving Therapy offered through a web platform

INTERVENTIONS:
Other: Problem Solving Therapy offered through a web platform — Problem Solving Therapy offered through a web platform. There will be four sessions, during the first four weeks of treatment, and subsequent sessions are dedicated to refining problem-solving skills. Participants set treatment goals; different ways to reach goals are discussed and evaluated; action plans are created, and its effectiveness is evaluated to achieve the objectives. Participants are expected to implement plans and apply the problem-solving model to additional problems between sessions. In the last two sessions, participants create a relapse prevention plan using the problem-solving therapy model.
  Arms: Problem Solving Therapy offered through a web platform
Other: Conventional web platform — The conventional web platform, which will contain the general content on stress coping techniques.
  Arms: Conventional web platform

SUMMARY:
Work-related stress is a problem due to its repercussions on workers' health and productivity, which is why workplace interventions are required to reduce stress levels through coping techniques. One of the interventions in mental health to reduce levels of work stress are those based on the Internet and mobile applications, with proven effectiveness. Among the interventions are cognitive-behavioral therapies and within these the Problem Solving Therapy (PST).

Therefore, there is a need to study the effect of Problem Solving Therapy offered through a web platform on the levels of self-perceived stress. However, there have been no studies on mental health interventions such as the TSP for the reduction of stress levels in office workers. For this reason, the objective of the study is to determine, through a randomized cluster trial, the effectiveness of problem-solving therapy offered through a web platform on self-perceived stress levels. Two scales will measure the levels of stress; one for self-perceived stress and another for work-related stress. Workers who have a high score on both scales will be enrolled. The establishments assigned to the intervention will receive the TSP distributed in 4 sessions. The establishments in the control group would have access to a web page with information on stress management. Immediately after having finished the last session, self-perceived stress levels will be evaluated. One month later a new measurement will be made to evaluate the persistence of the effect.

DETAILED DESCRIPTION:
The objective of the study is to determine, through a randomized cluster trial, the effectiveness of problem-solving therapy offered through a web platform on self-perceived stress levels.

Overall objective Evaluate the effect of Problem Solving Therapy offered through a web platform, on the self-perceived stress level of administrative workers.

Specific objectives

* Develop and validate a web platform with problem-solving therapy.
* Determine the cut-off point of self-perceived stress measurement scales.
* Evaluate the factors associated with stress in office workers.
* Compare the levels of Perceived stress scale (PSS) before and after the use of a web platform with educational material in Problem Solving Therapy (PST).
* Compare the effect of a conventional platform versus the Problem Solving Therapy offered through a web platform on self-perceived stress levels.
* Compare the levels of occupational stress (OSS) before and after the use of a web platform with educational material in Problem Solving Therapy (PST).
* Compare the effect of Problem Solving Therapy offered through a web platform versus a conventional web platform on work stress levels (WSS).
* Evaluate the correlation between the perceived stress scale and the occupational stress scale (OSS).

ELIGIBILITY:
Inclusion Criteria:

* Workers between 25 to 50 years of age poor conditions to be able to develop a therapy through a web platform.
* Workers with self-perceived stress scale and work stress with scores considered as stress.
* Working time ≥ one year.
* With signed informed consent.
* Workers with access to a computer connected to the internet during their working hours.
* Workers with ranges on the stress scale up to 2 standard deviations above the average.

Exclusion Criteria:

* Workers are taking anti-anxiety drugs and antidepressants, who scheduled their vacations during the follow-up period.
* People who for any physical or mental disability cannot use the web platform
* Workers with ranges on the stress scale for above three standard deviations above the average.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-09-28 (Estimated)

PRIMARY OUTCOMES:
Change in Self-perceived stress scale score | 0 and 5 weeks
  Perceived Stress Scale (PSS) It's formed by 14 items that measure the degree to which, during the last month, people have felt upset or worried or, on the contrary, have felt confident in their ability to control their personal problems. Scale scores between 0-56, with higher scores indicating greater stress perceived. Use a five-way Likert response format with a range of 0 "Never") to 4 ("Very often"). The cut point for determinate stress is 20.9 points (14 + 1 SD (6.9)) for hispanics. [ L. Harris Pol]

SECONDARY OUTCOMES:
Change in Occupational stress scale | 0 and 5 weeks
  Change in Occupational stress scale. This instrument has as author ILO-WHO. The questions are 25 with 7 alternatives such as answers ranging from the score from 1 to 7, of as follows.
  [1= if the condition 'Never' is a source of stress. 2 = if the condition 'Rarely' is a source of stress. 3 = if the condition 'Occasionally' is a source of stress 4 = if the condition 'Sometimes' is a source of stress. 5 = if the condition 'Frequently' is a source of stress 6 = if the condition "specifically" is a source of stress. 7 = if the "Always" condition is a source of stress.] The scale determinate the cut point for stress in 120 for Peruvian population. (Suaréz A. 2013)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Peruana Cayetano Heredia, Lima, Peru

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared

REFERENCES:
- [Background] Heber E, Ebert DD, Lehr D, Nobis S, Berking M, Riper H. Efficacy and cost-effectiveness of a web-based and mobile stress-management intervention for employees: design of a randomized controlled trial. BMC Public Health. 2013 Jul 15;13:655. doi: 10.1186/1471-2458-13-655. PMID 23855376
- [Result] Heber E, Lehr D, Ebert DD, Berking M, Riper H. Web-Based and Mobile Stress Management Intervention for Employees: A Randomized Controlled Trial. J Med Internet Res. 2016 Jan 27;18(1):e21. doi: 10.2196/jmir.5112. PMID 26818683